CLINICAL TRIAL: NCT04844528
Title: Randomized Phase 2 Studying the Effects of Nicotinamide in Patients With Chronic Lymphocytic Leukemia (CLL) With History of Non-melanoma Skin Cancers (NMSC)
Brief Title: Effects of Nicotinamide in Patients With Chronic Lymphocytic Leukemia With History of Non-melanoma Skin Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Huntsman Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HCI141430
Record Dates: First submitted 2021-04-12; First posted 2021-04-14 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukemia; Non-melanoma Skin Cancer (NMSC)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Niacinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotinamide, Then Nicotinamide (Experimental): Consenting patients with CLL who have had at least one NMSC diagnosed in the past year will be randomized to receive oral nicotinamide 500 mg twice daily (BID) for 1 year. Patients will be stratified according to CLL therapy and the number of prior NMSC. At the end of 1 year, patients will be unblinded, and all patients will receive Nicotinamide 500 mg BID for an additional year.
  Interventions: Drug: Nicotinamide
- Placebo, Then Nicotinamide (Experimental): Consenting patients with CLL who have had at least one NMSC diagnosed in the past year will be randomized to receive placebo twice daily (BID) for 1 year. Patients will be stratified according to CLL therapy and the number of prior NMSC. At the end of 1 year, patients will be unblinded, and all patients will receive Nicotinamide 500 mg BID for an additional year.
  Interventions: Drug: Nicotinamide; Drug: Placebo

INTERVENTIONS:
Drug: Nicotinamide — Oral nicotinamide 500 mg twice daily (BID).
  Other Names: Niacinamide
Drug: Placebo — Oral placebo twice daily for the first year.
  Arms: Placebo, Then Nicotinamide

SUMMARY:
This is a randomized, phase II, double-blind, placebo-controlled trial with planned crossover to the intervention arm after 1 year.

Consenting patients with CLL who have had at least one NMSC diagnosed in the past year will be randomized to receive either oral nicotinamide 500 mg twice daily (BID) for 1 year or oral placebo 1 tablet twice daily for 1 year. Patients will be stratified according to CLL therapy and the number of prior NMSC. At the end of 1 year, patients will undergo dermatologic examination and the number of new NMSC will be quantified. The number of patients who develop new NMSC in each arm will be documented. At this time, patients will be unblinded and all patients will receive Nicotinamide 500 mg BID for an additional year. At the end of this second year, patients will again undergo dermatologic examination, and the number of new NMSC will be quantified. The number of patients who develop NMSC will be documented. Skin biopsies will be taken for correlative studies.

Enrollment will be split into two parts separated by an interim analysis. Part 1 will accrue 40 patients: 20 to each arm. After 40 patients have completed their 12 month visit an interim futility analysis will be conducted prior to recruiting more patients. The study will stop if the difference in the number of patients with NMSC between control and treatment arms is 0 or less (i.e., absolutely no evidence that the treatment is better than control). If the trial is not stopped, the investigators will proceed with Part 2 and recruit 46 more patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged ≥ 18 years.
* Confirmed diagnosis of CLL or small lymphocytic leukemia (SLL) per iwCLL 2018 criteria.
* History of ≥1 non-melanoma skin cancer (NMSC) diagnosed within the last 5 years
* Adequate liver function as defined as:

  * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN)

    ---Subjects with a known diagnosis of Gilbert's Syndrome: direct bilirubin ≤ 1.5x ULN
  * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN
* For female subjects: Negative pregnancy test or evidence of post-menopausal status. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  --Women < 50 years of age:
  * Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and
  * Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution; or
  * Underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
* Women ≥ 50 years of age:

  * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments; or
  * Had radiation-induced menopause with last menses >1 year ago; or
  * Had chemotherapy-induced menopause with last menses >1 year ago; or
  * Underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
* Female subjects of childbearing potential and male subjects with a sexual partner of childbearing potential must agree to use a highly effective method of contraception.

Exclusion Criteria:

* Received cytotoxic chemotherapy (including fludarabine, cyclophosphamide, bendamustine, or chlorambucil) within the last 6 months
* Received allogeneic stem cell transplant within the last 6 months.
* Taking nicotinamide or niacin supplements within the last 4 weeks.
* Taken acitretin or other oral retinoids within the past 6 months
* Received field treatment for AKs (topical use of 5-fluorouracil, imiquimod, diclofenac, retinoids; topical photodynamic therapy for AKs; laser resurfacing or chemical peel treatments for AKs) within the previous 4 weeks
* Large areas of confluent skin cancer at baseline preventing accurate assessment and counting of individual new skin cancers
* Need for ongoing carbamazepine use (possible interaction with nicotinamide)
* Severe GI malabsorption that may interfere with absorption of nicotinamide (per investigator's discretion)
* Patients with an expected life expectancy < 2 years
* Current evidence of uncontrolled, diabetes.
* Current evidence or history of peptic ulcer disease.
* Known HIV infection with a detectable viral load within 6 months of the anticipated start of treatment.

Note: Subjects on effective antiretroviral therapy with an undetectable viral load within 6 months of the anticipated start of treatment are eligible for this trial.

* Known active uncontrolled infection.
* Medical, psychiatric, cognitive, or other conditions that may compromise the subject's ability to understand the subject information, give informed consent, comply with the study protocol or complete the study.
* Known prior severe hypersensitivity to investigational product (IP) or any component in its formulations (NCI CTCAE v5.0 Grade ≥ 3).
* Subjects taking prohibited medications as described in study protocol. A washout period of prohibited medications for a period of at least five half-lives or as clinically indicated should occur before the start of treatment.
* Have ever received a solid organ transplant and are currently taking immunosuppressive medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of CLL patients who develop a new NMSC after 1 year of nicotinamide therapy. | 1 year
  evaluate whether nicotinamide can reduce the number of patients who develop one or more new NMSC versus placebo in CLL patients with a history of NMSC.

SECONDARY OUTCOMES:
Number of new NMSC on skin exam after 1 year of treatment | 1 year
  assess the effect of oral nicotinamide on the number of new NMSC in patients with CLL who have previously been diagnosed with a NMSC.
proportion of CLL patients who develop squamous cell carcinoma (SCC) on skin exam after 1 and 2 years of treatment. | up to 2 years
  assess whether nicotinamide can reduce the number of patients who develop a SCC versus placebo in CLL patients with a history of NMSC.
proportion of CLL patients who develop basal cell carcinoma (BCC) on skin exam after 1 and 2 years of treatment. | up to 2 years
  assess whether nicotinamide can reduce the number of subjects who develop a BCC versus placebo in CLL patients with a history of NMSC
proportion of CLL patients who develop actinic keratosis (AK) on skin exam after 1 and 2 years of treatment. | up to 2 years
  evaluate whether nicotinamide can reduce the number of subjects who develop AK versus placebo in CLL patients with a history of NMSC
number of new NMSC developed during year 1 and year 2 for patients who receive placebo during the first year | 2 years
  evaluate whether nicotinamide can reduce the number of recurrent NMSC in the same patient between year 1 on placebo therapy and year 2 on nicotinamide therapy
objective response rate (the proportion of subjects achieving a complete response [CR] or partial response [PR]) and complete response rate as calculated per International Workshop on CLL (IWCLL) 2018 Criteria at Month 6, 12, 18, and 24 | up to 24 months
  2.2.6 To compare objective response rates (CR + PR) and CR rates between patients not on active CLL therapy who receive nicotinamide versus placebo
objective response rate (the proportion of subjects achieving a CR or PR) and complete response rate as calculated per International Workshop on CLL (IWCLL) 2018 Criteria at Month 6, 12, 18, and 24 | up to 24 months
  2.2.7 To compare overall response rates (CR+ partial PR) and CR rates between patients not on active CLL therapy with and without mutations with DNA mismatch repair who receive nicotinamide versus placebo
frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by type, severity (as defined by the NIH CTCAE, version 5.0 and iwCLL), seriousness, duration, and relationship to study treatment | up to 24 months
  evaluate the safety and tolerability of each arm

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Fitzgerald, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Royle JA, Baade PD, Joske D, Girschik J, Fritschi L. Second cancer incidence and cancer mortality among chronic lymphocytic leukaemia patients: a population-based study. Br J Cancer. 2011 Sep 27;105(7):1076-81. doi: 10.1038/bjc.2011.313. Epub 2011 Aug 16. PMID 21847118
- [Background] Kleinstern G, Rishi A, Achenbach SJ, Chaffee KR, Kay NE, Shanafelt TD, et al. Skin Cancers Among Chronic Lymphocytic Leukemia (CLL) Patients - the Effect of UV Radiation and CLL Clinical Characteristics. Blood. 2016;128(22):4772-.
- [Background] Mehrany K, Weenig RH, Pittelkow MR, Roenigk RK, Otley CC. High recurrence rates of squamous cell carcinoma after Mohs' surgery in patients with chronic lymphocytic leukemia. Dermatol Surg. 2005 Jan;31(1):38-42; discussion 42. doi: 10.1111/j.1524-4725.2005.31006. PMID 15720094
- [Background] Mehrany K, Weenig RH, Lee KK, Pittelkow MR, Otley CC. Increased metastasis and mortality from cutaneous squamous cell carcinoma in patients with chronic lymphocytic leukemia. J Am Acad Dermatol. 2005 Dec;53(6):1067-71. doi: 10.1016/j.jaad.2005.08.055. PMID 16310071
- [Background] Chen AC, Martin AJ, Choy B, Fernandez-Penas P, Dalziell RA, McKenzie CA, Scolyer RA, Dhillon HM, Vardy JL, Kricker A, St George G, Chinniah N, Halliday GM, Damian DL. A Phase 3 Randomized Trial of Nicotinamide for Skin-Cancer Chemoprevention. N Engl J Med. 2015 Oct 22;373(17):1618-26. doi: 10.1056/NEJMoa1506197. PMID 26488693
- [Background] Hampras SS, Locke FL, Chavez JC, Patel NS, Giuliano AR, Miller K, Gheit T, Tommasino M, Rollison DE. Prevalence of cutaneous viral infections in incident cutaneous squamous cell carcinoma detected among chronic lymphocytic leukemia and hematopoietic stem cell transplant patients. Leuk Lymphoma. 2018 Apr;59(4):911-917. doi: 10.1080/10428194.2017.1342822. Epub 2017 Jul 6. PMID 28679298
- [Background] Park J, Halliday GM, Surjana D, Damian DL. Nicotinamide prevents ultraviolet radiation-induced cellular energy loss. Photochem Photobiol. 2010 Jul-Aug;86(4):942-8. doi: 10.1111/j.1751-1097.2010.00746.x. Epub 2010 May 13. PMID 20492562
- [Background] Yiasemides E, Sivapirabu G, Halliday GM, Park J, Damian DL. Oral nicotinamide protects against ultraviolet radiation-induced immunosuppression in humans. Carcinogenesis. 2009 Jan;30(1):101-5. doi: 10.1093/carcin/bgn248. Epub 2008 Nov 20. PMID 19028705
- [Background] Surjana D, Halliday GM, Martin AJ, Moloney FJ, Damian DL. Oral nicotinamide reduces actinic keratoses in phase II double-blinded randomized controlled trials. J Invest Dermatol. 2012 May;132(5):1497-500. doi: 10.1038/jid.2011.459. Epub 2012 Feb 2. No abstract available. PMID 22297641
- [Background] Knip M, Douek IF, Moore WP, Gillmor HA, McLean AE, Bingley PJ, Gale EA; European Nicotinamide Diabetes Intervention Trial Group. Safety of high-dose nicotinamide: a review. Diabetologia. 2000 Nov;43(11):1337-45. doi: 10.1007/s001250051536. PMID 11126400
- [Background] Niren NM. Pharmacologic doses of nicotinamide in the treatment of inflammatory skin conditions: a review. Cutis. 2006 Jan;77(1 Suppl):11-6. PMID 16871774
- [Background] Lampeter EF, Klinghammer A, Scherbaum WA, Heinze E, Haastert B, Giani G, Kolb H. The Deutsche Nicotinamide Intervention Study: an attempt to prevent type 1 diabetes. DENIS Group. Diabetes. 1998 Jun;47(6):980-4. doi: 10.2337/diabetes.47.6.980. PMID 9604880
- [Background] PubChem Compound Summary for CID 936, Nicotinamide: National Center for Biotechnology Information; [Available from: https://pubchem.ncbi.nlm.nih.gov/compound/Nicotinamide.
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Glanz K, Yaroch AL, Dancel M, Saraiya M, Crane LA, Buller DB, Manne S, O'Riordan DL, Heckman CJ, Hay J, Robinson JK. Measures of sun exposure and sun protection practices for behavioral and epidemiologic research. Arch Dermatol. 2008 Feb;144(2):217-22. doi: 10.1001/archdermatol.2007.46. PMID 18283179
- [Background] Rai KR, Sawitsky A, Cronkite EP, Chanana AD, Levy RN, Pasternack BS. Clinical staging of chronic lymphocytic leukemia. Blood. 1975 Aug;46(2):219-34. PMID 1139039
- [Background] International CLL-IPI working group. An international prognostic index for patients with chronic lymphocytic leukaemia (CLL-IPI): a meta-analysis of individual patient data. Lancet Oncol. 2016 Jun;17(6):779-790. doi: 10.1016/S1470-2045(16)30029-8. Epub 2016 May 13. PMID 27185642